CLINICAL TRIAL: NCT05752110
Title: Does Subanesthetic Dose of Ketamine Given at Induction of Anesthesia Improve Postoperative Mood In Women Undergoing Fractional Curettage? A Randomized Controlled Trial
Brief Title: Effects of Subanesthetic Dose of Ketamine Given on Postoperative Mood in Patients Undergoing Fractional Curettage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sevim Baltali, Principal Investigator; M.D. Department of Anesthesiology, Istanbul Training and Research Hospital, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 106/2022
Record Dates: First submitted 2023-02-10; First posted 2023-03-02 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Ketamine; Minor Surgical Procedure; Total Mood Score; Woman
Keywords: ketamine; POMS questionnary; acute Mood; fractional curettage; propofol
MeSH Terms: interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Active Comparator): Received 0.5mg/kg IV single dose ketamine in addition to propofol and fentanyl anesthesia at induction period of anesthesia.
  Interventions: Drug: Ketamine
- Control (Placebo Comparator): Received 0.05ml/kg IV % 0.9 saline in addition to propofol and fentanyl anesthesia at induction period of anesthesia.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ketamine — 0,5mg/kg single dose Ketamine (0.05ml/kg) intravenously administered
  Other Names: subanesthetic dose of Ketamine
  Arms: Ketamine
Other: Saline — 0.09% Saline (0.05ml/kg) intravenously administered
  Other Names: Placebo
  Arms: Control

SUMMARY:
When given intravenously in doses below 1.2mg/kg, ketamine has been shown to work as an antidepressant. Ketamine is a common induction drug used during general anesthesia. It is known to reduce postoperative pain in this instance. Limited studies have evaluated the effect of a single subanesthetic dosage of ketamine administered as an adjunct to general anesthesia on acute mood states in patients undergoing minor surgery. The aim of this randomized controlled study was to examine if a single intravenous administration of 0.5 mg/kg ketamine given at the induction of propofol/fentanyl anesthesia has an effect on acute mood states before the discharge of women undergoing fractional curettage.

DETAILED DESCRIPTION:
Women admitted for fractional curettage between the ages of 18 and 75 were asked if they would like to participate in the study. Exclusion criteria included uncontrolled hypertension, pregnancy, history of psychologic disorders, use of brain-affecting medicines, substance abuse, seizure disorders, or ketamine allergy. After receiving informed consent, the patient would be given a POMS questionnaire. The participants were then assigned randomly to one of two groups. Group A will receive ketamine intravenously at a dose of 0.5 mg/kg as part of the induction process for general anesthesia. In addition to their anesthetic, Group B will get the same amount of saline instead of ketamine. Patients were treated by a different anesthetic professional (who is blinded to the group the patient is in). All other induction medicines were administered at the discretion of the anesthesiologist. Two hours after the surgery, participants were again administered the POMS questionnaire, questioned about their pain level, and their data sheet was updated accordingly. During the trial, the levels of sedation, systolic and diastolic blood pressures and heart rate were measured. In addition, any adverse events were documented.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients (>18 years) undergoing fractional curettage

Exclusion Criteria:

* American Society of Anesthesiologists' physical status ≥ 3
* History of psychological disorders
* Use of drugs affect central nervous system
* Substance abuse
* Chronic pain
* Pregnancy
* Seizure disorders
* Cardiovascular, hepatic or renal disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Comparing total mood scores of both groups using Profile of Mood States (POMS) Questionnaire. | Total Mood Score measured 120 minutes after surgery
  The Turkish version of Profile of Mood States (POMS) is an validated instrument that measures mood using a 58-item questionnaire with each item rated using a response scale of five categories ranging from "not at all" to "very strong". Higher score indicates worse mood.As a global measure of affective state, a total mood score (TMS) is calculated by combining the negative mood subscore (NMS) totals (fatigue-inertia, anger-hostility, confusion-bewilderment, depression-dejection, tension-anxiety,) and subtracting the positive mood subscore (PMS) (vigor-activity). The minimum value of TMS is -24, the maximum value is+177.
Impact of clinical variables on total mood scores using Profile of Mood States (POMS) | 120 minutes after surgery
  We perform multiple linear regression analyses to examine the independent predictors of changes in postoperative TMS in the entire study group, patients in group-K and group-C, separately. Postoperative TMS is the dependent variable; menopausal status, parity, educational level, body mass index (BMI) and preoperative TMS are independent variables.

SECONDARY OUTCOMES:
Numeric rating scale for pain assessment | 120 minutes after surgery
  Numeric rating scale score (NRS) is commonly used for measuring pain intensity. It is scored from 0-10; 0 means no pain and 10 is the worst pain imaginable. NRS assessed at the 120 minutes postoperatively
Systolic blood pressure | immediately before surgery and 120 minutes after surgery
  Measuring systolic blood pressure (mmHg) before surgery and 120 minutes after surgery and comparing values between and within group K and group C
diastolic blood pressure | immediately before surgery and 120 minutes after surgery
  Measuring diastolic blood pressure (mmHg) before surgery and 120 minutes after surgery and comparing values within groups and comparing values between and within group K and group C
heart rate | immediately before surgery and 120 minutes after surgery
  Measuring number of heart beats per minute before surgery and 120 minutes after surgery and comparing values within groups and comparing values between and within group K and group C
The Michigan Sedation Score assessment | immediately Before surgery, 60 minutes after surgery and 120 minutes after surgery
  Comparing depth of sedations of two groups using the University of Michigan Sedation Scale (UMSS). This sedation scale ranges from zero to four with higher numbers indicating deeper sedation.
Diplopia | 120 minutes after surgery
  Presence of absence of diplopia reported in clinical records electronic database by nurse or physician within time frame
Headache | 120 minutes after surgery
  Presence of absence of headache reported in clinical records electronic database by nurse or physician within time frame
Psychedelic phenomena | 120 minutes after surgery
  Presence of absence of psychedelic phenomena reported in clinical records electronic database by nurse or physician within time frame
Nausea | 120 minutes after surgery
  Presence of absence of nausea reported in clinical records electronic database by nurse or physician within time frame
Vomiting | 120 minutes after surgery
  Presence of absence of vomiting reported in clinical records electronic database by nurse or physician within time frame
Patient satisfaction | 120 minutes after surgery
  Evaluation of patient satisfaction 120 minutes after surgery. Satisfaction is rated on a scale of 1 to 4 (1 perfect, 2 good, 3 moderate, and 4 bad).
Physician satisfaction | 120 minutes after surgery
  Evaluation of physician satisfaction 120 minutes after surgery. Satisfaction is rated on a scale of 1 to 4 (1 perfect, 2 good, 3 moderate, and 4 bad).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet TOPTAS, Ass.Prof.Dr, Study Chair — Istanbul Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Training and Research Hospital, Istanbul, Fatih
  - IstanbulTRH, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baltali S, Ciftci E, Baltali M, Haliloglu M, Ercan A, Tunay A, Celik Z, Bozay B, Toptas M. Ketamine's impact on mood after day-case surgery and its relation to obesity: a randomised controlled trial in women undergoing fractional curettage. BMC Womens Health. 2025 Jul 30;25(1):380. doi: 10.1186/s12905-025-03920-y. PMID 40739637